CLINICAL TRIAL: NCT03935490
Title: The Transrectus Sheath Pre-peritoneal (TREPP) Technique for Strangulated Inguinal Hernia: a Case-series
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: St Jansdal Hospital (Other)
Responsible Party: Principal Investigator, Thomas Zwols, Principal Investigator, University Medical Center Groningen
Other Study IDs: 201900143
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Strangulated Inguinal Hernia
Keywords: Inguinal hernia; Strangulated; TREPP; Transrectus sheath pre-peritoneal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- e-TREPP: Patients with strangulated inguinal hernia treated with e-TREPP
  Interventions: Procedure: emergency transrectus sheath pre-peritoneal mesh repair (e-TREPP)

INTERVENTIONS:
Procedure: emergency transrectus sheath pre-peritoneal mesh repair (e-TREPP) — The Trans REctussheath PrePeritoneal mesh repair (TREPP) was developed in 2006 as an open preperitoneal technique to reduce CPIP. In short: a 4-5 centimeters (cm) transverse incision is made about 1 cm above the localization of the deep inguinal ring. The anterior rectus sheath is opened. After retracting the rectus muscle medially, the preperitoneal space (PPS) is bluntly dissected and a complete overview can be achieved. All possible hernia orifices can be visualized such as: a direct, indirect, pantaloon, and/or femoral hernia. A self-expandable mesh is then positioned in the PPS. Due to the "upstream principle" no mesh fixation is necessary.

SUMMARY:
n the Sint Jansdal Hospital in Harderwijk, the Netherlands, the TREPP technique is the standard operating procedure for patients with inguinal hernia. Starting from 2006, this procedure has also been used on patients that presented with an acute strangulated inguinal hernia in the emergency department, instead of the more common Lichtenstein technique. The goal of this retrospective case series is to assess the feasibility of the TREPP technique in case of an acute strangulated inguinal hernia. Patient records from 2006 until 2016 will be used to search for patients treated for acute inguinal hernia in that period. After applying the in- and exclusion criteria, patients who are eligible for inclusion will be contacted by telephone. They will be asked if they are willing to visit the surgical outpatient department once and fill out two questionnaires. The data of these questionnaires will be analyzed and published.

ELIGIBILITY:
Inclusion Criteria:

* Emergency surgery for suspected strangulated inguinal hernia (within 6 hours after admission)
* e-TREPP performed

Exclusion Criteria:

* No emergency surgery (for instance, surgery day after admission or later).
* No e-TREPP performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From all acute inguinal hernia repairs patient records will searched for e-TREPP procedures. All patients will be asked to visit the outpatient department.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Chronic postoperative inguinal pain according to Visual Analog Scale | From surgery date up to 12 years postoperatively
  Patients will be asked to fill out the VAS on a horizontal line of 10 millimeters long. Patients will be asked to mark the point that indicated the amount of pain they experience. The distance from the left marker will be measured, with increasing distance at greater pain intensity.
Recurrence rate | From surgery date up to 12 years postoperatively
  Patient electronic records will be searched for re-operations for recurrent inguinal hernia. Also, patients will be asked in the outpatient department if they received recurrence surgery or suffer new complaints.

SECONDARY OUTCOMES:
Short-term complications | Complications occuring from the start of the operation up to 30 days postoperative
  Short term complications included: hematoma, wound infection, re-admission rate, medical complications and death. These complications will be retrospectively analyzed via the electronic patient files. They will be verified at the outpatient department.
Sexual complaints related to e-TREPP | Between >30 days postoperatively and through study completion, average 6 years
  All patients will be asked if they experienced any sexual problems related to the e-TREPP surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- St Jansdal Hospital, Harderwijk, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No